CLINICAL TRIAL: NCT06611475
Title: Prediction of MMSE Scores for Cognitive Impairment: A Machine Learning Analysis of Oral Health and Demographic Data in Individuals Over 60 Years of Age
Brief Title: Prediction of MMSE Scores for Cognitive Impairment
Status: Completed | Type: Observational
Sponsor: Blekinge Institute of Technology (Other)
Responsible Party: Sponsor
Other Study IDs: BTH-6.1.1-0156-2024
Record Dates: First submitted 2024-09-17; First posted 2024-09-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-09

CONDITIONS: Cognitive Impairment; Healthy Control
Keywords: Classification; Machine Learning; Mini-Mental State Examination; Cognitive Impairment; Oral Health
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MMSE ≤26: 339 participants
  Interventions: Other: MMSE ≤26
- MMSE 30: 354 participants
  Interventions: Other: MMSE ≤26

INTERVENTIONS:
Other: MMSE ≤26 — A dataset comprising participants with MMSE scores of ≤26 and 30 will be used to evaluate the classification performance of various machine learning techniques.
  Other Names: MMSE 30

SUMMARY:
This study aims to explore the potential of using machine learning (ML) algorithms to predict cognitive status, specifically MMSE scores, based on oral health and demographic data. The objective is to evaluate the effectiveness of various ML models and identify the most relevant oral health indicators for predicting MMSE scores of 30 (normal cognition) or ≤26 (cognitive impairment) in individuals aged 60 and above.

DETAILED DESCRIPTION:
This cross-sectional study utilizes oral health and demographic data from two existing cohort studies: the European collaborative study Support Monitoring and Reminder Technology for Mild Dementia (SMART4MD) and the Swedish National Study on Aging and Care (SNAC-B). Participants aged 60 years or older will be included in the analysis. The data will be used to develop and evaluate machine learning models for predicting cognitive status.

Objectives:

1. Primary Objective: To assess the potential of oral health parameters for binary classification of MMSE scores (30 vs. ≤26).
2. Secondary Objective: To identify the most influential oral health parameters contributing to cognitive impairment predictions.
3. Tertiary Objective: To compare the performance of Random Forest (RF), Support Vector Machine (SVM), and CatBoost (CB) classifiers in predicting MMSE scores using oral health data.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 60 years or older.
* Participants with recorded oral health parameters and MMSE scores of either 30 or ≤26.

Exclusion Criteria:

* Individuals with MMSE scores of 27, 28, or 29, as these scores represent a transition phase between normal cognition and cognitive impairment, which could introduce variability.
* Individuals younger than 60 years.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Data collected from the European collaborative study Support Monitoring and Reminder Technology for Mild Dementia (SMART4MD) and the Swedish National Study on Aging and Care (SNAC-B) will be analyzed. Participants aged 60 years or older will be included in the analysis.
Sampling Method: Non-Probability Sample
Enrollment: 693 (Actual)
Dates: Start 2024-06-10 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-11-10 (Actual)

PRIMARY OUTCOMES:
Detection perfomance | 5 mounths
  The study measures the classification performance of Machine Learning classifiers. Performance metrics, Accuracy, precision, recall, F1-Score and confusion matrix will be used for the evaluation. The examination of the most important features relied on SHAP summary plots, providing visualizations of the influence of parameter groups on the output, organized by their importance. This importance is based on SHAP values, offering insights into features' effects on the ML model's decision-making process

CONTACTS AND LOCATIONS:
Locations (1):
- Blekinge institute of Technology, Karlskrona, Sweden

IPD SHARING:
Plan to Share IPD: No
Participant data can not be shared due to the GDPR.